CLINICAL TRIAL: NCT05704517
Title: Progressive Familial Intrahepatic Cholestasis in Indian Children - Establishing an Indian PFIC Registry
Status: Recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Collaborators: Apollo Hospital, New Delhi, India (Other); Sahyadri Superspeciality Hospital Pvt Ltd, Pune (Unknown); Glenegales Global Health City, Chennai (Unknown); KEM Hospital Research Centre (Other); Jaslok Hospital and Research Centre (Other); Institute of Child Health, Chennai (Unknown)
Responsible Party: Sponsor
Other Study IDs: India_PFIC
Record Dates: First submitted 2022-12-21; First posted 2023-01-30 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Progressive Familial Intrahepatic Cholestasis
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project will amalgamate data from several large Indian centers to describe the genotype, clinical spectrum, natural course, genotype-phenotype correlation, outcome, and response to medical therapy in Indian children with progressive familial intrahepatic cholestasis (PFIC). This will be the first such Indian registry of children with PFIC. There are currently limited single-center studies describing the genotype, natural course, and outcome of Indian children with PFIC.

Data will be collected retrospectively from the participating centers across the country. Only genetically confirmed cases would be included.

DETAILED DESCRIPTION:
There is a lack of robust literature from India on PFIC. The study would be the first to extensively describe the genotype of Indian children with PFIC and their natural course. Being a multicentric study, the results generated would therefore be applicable to the whole of the country. Understanding the prevalent genotypes in the Indian population and their related phenotype would help both the individual management decisions of these patients and further policy-making for their diagnosis and treatment. With the advent of genetic diagnosis through sequencing techniques and these tests becoming more affordable, every Indian center is now diagnosing a fair number of these cases which used to go undiagnosed previously. This has changed the landscape of cholestatic liver disease in children where PFICs are now the most prevalent pediatric cholestatic disorder. European studies have demonstrated 2 common mutations where patients respond very well to surgical biliary diversion and have good native liver survival. These mutations have rarely been reported in India. Results from this study could thus guide appropriate decision-making based on outcome and help choose the modality of treatment for the individual patient - medical, surgical biliary diversion, or liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Genetically proven homozygous or compound heterozygous mutations of ATP8B1/ ABCB11/ ABCB4/ TJP2/ NR1H4/ MYO5B/ USP53/ KIF12 AND
* Clinical and biochemical evidence of chronic cholestatic disease AND / OR
* Histological features of intrahepatic cholestasis with suggestive immunohistochemistry

Exclusion Criteria:

* Genetic analysis showing mutations unrelated to intrahepatic cholestasis according to database
* Clinical, biochemical, and histological evidence of progressive familial intrahepatic cholestasis without a genetic sequencing report

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All genetically confirmed cases of progressive familial intrahepatic cholestasis (PFIC)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Native liver survival (in percentage) at the latest follow up in different types of PFIC | Through study completion - average of 1 year
  The proportion of patients of each subtype of PFIC who have survived with their own with their native liver till the time of last follow up

SECONDARY OUTCOMES:
Describe the spectrum of genetic mutations in Indian children with familial intrahepatic cholestasis | Through study completion - average of 1 year
  This objective would be assessed by studying the frequency of each of these subtypes of PFIC and describing the various genotypes under each subtype.
Genotype-phenotype correlation in Indian children with various types of progressive familial intrahepatic cholestasis | Through study completion - average of 1 year
  Well defined clinical parameters (jaundice, pruritus, presentation, presence of cirrhosis) and clinical end points (death, liver transplantation, native liver survival) would be used to describe the genotype-phenotype correlation. We will try to club various mutations into categories based on the type of mutations to better assess the genotype-phenotype correlation.
Analyse the natural course after surgical biliary diversion in Indian children with various types of progressive familial intrahepatic cholestasis | Through study completion - average of 1 year
  We will analyze the response to surgical biliary diversion in various types of PFIC with emphasis on identifying the genotypes likely to gain maximum benefit through this procedure. Biochemical parameters to assess/ predict the response would be evaluated by regression analysis.
Complications after liver transplantation in children with various types of progressive familial intrahepatic cholestasis till the time of last follow up | Through study completion - average of 1 year
  The proportion of children going for liver transplantation at various time points would be assessed. Genetic, clinical or biochemical parameters predicting need for imminent/ future liver transplantation would be determined by regression analysis.
Proportion of patients surviving with native liver in uncommon variants of progressive familial intrahepatic cholestasis | Through study completion - average of 1 year
  Describe the prevalence, natural course and outcome of uncommon variants of progressive familial intrahepatic cholestasis in Indian children
Develop and maintain a registry of Indian patients with progressive familial intrahepatic cholestasis (Indian PFIC registry) | Through study completion - average of 2 years
  A registry (Indian PFIC registry) would be maintained with use of appropriate data managing software.

CONTACTS AND LOCATIONS:
Overall Officials: Bikrant B Lal, MD, DM, Principal Investigator — Institute of Liver and Biliary Sciences, New Delhi
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: No
Individual patient data would not be shared with other researchers.

REFERENCES:
- [Background] Agarwal S, Lal BB, Rawat D, Rastogi A, Bharathy KG, Alam S. Progressive Familial Intrahepatic Cholestasis (PFIC) in Indian Children: Clinical Spectrum and Outcome. J Clin Exp Hepatol. 2016 Sep;6(3):203-208. doi: 10.1016/j.jceh.2016.05.003. Epub 2016 May 24. PMID 27746616
- [Background] Sharma A, Poddar U, Agnihotry S, Phadke SR, Yachha SK, Aggarwal R. Spectrum of genomic variations in Indian patients with progressive familial intrahepatic cholestasis. BMC Gastroenterol. 2018 Jul 4;18(1):107. doi: 10.1186/s12876-018-0835-6. PMID 29973134
- [Background] Mitra S, Das A, Thapa B, Kumar Vasishta R. Phenotype-Genotype Correlation of North Indian Progressive Familial Intrahepatic Cholestasis type2 Children Shows p.Val444Ala and p.Asn591Ser Variants and Retained BSEP Expression. Fetal Pediatr Pathol. 2020 Apr;39(2):107-123. doi: 10.1080/15513815.2019.1641860. Epub 2019 Jul 23. PMID 31335238
- [Background] van Wessel DBE, Thompson RJ, Gonzales E, Jankowska I, Sokal E, Grammatikopoulos T, Kadaristiana A, Jacquemin E, Spraul A, Lipinski P, Czubkowski P, Rock N, Shagrani M, Broering D, Algoufi T, Mazhar N, Nicastro E, Kelly DA, Nebbia G, Arnell H, Bjorn Fischler, Hulscher JBF, Serranti D, Arikan C, Polat E, Debray D, Lacaille F, Goncalves C, Hierro L, Munoz Bartolo G, Mozer-Glassberg Y, Azaz A, Brecelj J, Dezsofi A, Calvo PL, Grabhorn E, Sturm E, van der Woerd WJ, Kamath BM, Wang JS, Li L, Durmaz O, Onal Z, Bunt TMG, Hansen BE, Verkade HJ; NAtural course and Prognosis of PFIC and Effect of biliary Diversion (NAPPED) consortium. Genotype correlates with the natural history of severe bile salt export pump deficiency. J Hepatol. 2020 Jul;73(1):84-93. doi: 10.1016/j.jhep.2020.02.007. Epub 2020 Feb 20. PMID 32087350
- [Background] van Wessel DBE, Thompson RJ, Gonzales E, Jankowska I, Shneider BL, Sokal E, Grammatikopoulos T, Kadaristiana A, Jacquemin E, Spraul A, Lipinski P, Czubkowski P, Rock N, Shagrani M, Broering D, Algoufi T, Mazhar N, Nicastro E, Kelly D, Nebbia G, Arnell H, Fischler B, Hulscher JBF, Serranti D, Arikan C, Debray D, Lacaille F, Goncalves C, Hierro L, Munoz Bartolo G, Mozer-Glassberg Y, Azaz A, Brecelj J, Dezsofi A, Luigi Calvo P, Krebs-Schmitt D, Hartleif S, van der Woerd WL, Wang JS, Li LT, Durmaz O, Kerkar N, Horby Jorgensen M, Fischer R, Jimenez-Rivera C, Alam S, Cananzi M, Laverdure N, Targa Ferreira C, Ordonez F, Wang H, Sency V, Mo Kim K, Chen HL, Carvalho E, Fabre A, Quintero Bernabeu J, Alonso EM, Sokol RJ, Suchy FJ, Loomes KM, McKiernan PJ, Rosenthal P, Turmelle Y, Rao GS, Horslen S, Kamath BM, Rogalidou M, Karnsakul WW, Hansen B, Verkade HJ; Natural Course and Prognosis of PFIC and Effect of Biliary Diversion Consortium. Impact of Genotype, Serum Bile Acids, and Surgical Biliary Diversion on Native Liver Survival in FIC1 Deficiency. Hepatology. 2021 Aug;74(2):892-906. doi: 10.1002/hep.31787. Epub 2021 Jul 13. PMID 33666275
- [Background] Alam S, Lal BB. Recent updates on progressive familial intrahepatic cholestasis types 1, 2 and 3: Outcome and therapeutic strategies. World J Hepatol. 2022 Jan 27;14(1):98-118. doi: 10.4254/wjh.v14.i1.98. PMID 35126842